CLINICAL TRIAL: NCT03864549
Title: The Effect of Oral Probiotics on Glycemic Control of Women With Gestational Diabetes Mellitus - Randomized, Double Blind, Placebo Controlled Trial, Phase 4
Brief Title: The Effect of Oral Probiotics on Glycemic Control of Women With Gestational Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0003-19
Record Dates: First submitted 2019-01-21; First posted 2019-03-06 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotic femina II (Experimental): research group will receive the probiotic formula Femina II (2 capsules/day) until delivery.
  Interventions: Dietary Supplement: Femina II
- Placebo (Placebo Comparator): control group will receive a placebo (2 capsules/day) until delivery.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Femina II — 2 capsules per day until delivery
  Arms: probiotic femina II
Other: Placebo — 2 capsules per day until delivery
  Arms: Placebo

SUMMARY:
Scientific background: Uncontrolled gestational diabetes mellitus (GDM) is associated with severe maternal and neonatal morbidities. Treatment of GDM is multidisciplinary and includes lifestyle changes and medications. However, the efficacy of these treatments is limited due to poor motivation, daily painful blood tests and multiple injections.

Probiotic supplements were shown to modulate the gut microbiome by reducing the adverse metabolic effects associated with pathogenic microbial colonization. Promising effects on glycemic control and insulin resistance in non-pregnant diabetic patients were reported. However, the effect of probiotics on glycemic control in GDM has not been elucidated.

Objectives: To examine the effect of a mixture of probiotic strains given daily on maternal glycemic parameters, and pregnancy outcomes among women with GDM.

Working hypothesis: Oral administration of probiotics will be effective in glucose control of patients with GDM and their neonates without causing significant adverse effects.

Type of research and methods of data collection: A prospective randomized, double blind, placebo controlled trial. Women newly diagnosed with GDM will be recruited and followed in the GDM clinic and Maternal-Fetal Medicine ward (including the research clinic) at Emek Medical Center. They will be divided into a research group, receiving the probiotic formula Femina II and a control group, receiving a placebo (2 capsules/day) until delivery. Glycemic control will be evaluated by daily glucose charts. After 2 weeks of diet and probiotic/placebo treatment and thereafter, pharmacotherapy will be started in case of poor glycemic control according to the daily glucose charts. Blood tests for glycated molecules will be performed. Fetal well-being and growth will be assessed. The primary outcomes are:

1. The rate of women requiring medications for glycemic control
2. Mean value of the mean daily glucose charts after 2 weeks of treatment with the study products.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who were diagnosed with GDM from 13 to 32.6 gestational weeks
* 18 years old and older
* Singleton pregnancy

Exclusion Criteria:

* Women with pre-gestational diabetes mellitus
* GDM diagnosed ≥ 33 gestational weeks
* Women using prophylactic antimicrobial treatment
* Immunocompromised women
* Multiple pregnancy
* Women taking oral probiotic products who refuse to stop the consumption (food-containing probiotics is not considered an exclusion criterion).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
The rate of women who will require pharmacotherapy for glycemic control. | During the length of pregnancy (up to 9 months)
Mean value of the mean daily glucose charts after 2 weeks of treatment with the study products. | 2 weeks

SECONDARY OUTCOMES:
The rate of women with controlled diabetes | During the length of pregnancy (up to 9 months)
Mean daily glucose charts | During the length of pregnancy (up to 9 months)
Mean daily pre-prandial glucose values | During the length of pregnancy (up to 9 months)
Mean daily post-prandial glucose values | During the length of pregnancy (up to 9 months)
Level of glycated molecules | During the length of pregnancy (up to 9 months)
The rate of women with mean pre-prandial values ≥ 95 mg/dl, mean post-prandial values ≥ 130 mg/dl, and mean daily glucose > 100 mg/dl | During the length of pregnancy (up to 9 months)
The rate of cesarean deliveries | At delivery
The rate of labor inductions | At delivery
The rate of birth weight≥4000 gr | At delivery
The rate of birth weight> 90th percentile | At delivery
The rate of admission to the neonatal intensive care unit | Within a week from delivery
Apgar score at 1 and 5 minutes from birth | Within 1-5 minutes after delivery
The rate of neonatal hypoglycemia | Within 1-2 days after delivery
The rate of neonatal hyperbilirubinemia | Within a week from delivery
The rate of neonatal polycythemia | Within a week from delivery
The rate of neonatal hypocalcemia | Within a week from delivery
The rate of neonatal hypomagnesemia | Within a week from delivery
Cord blood pH levels | At delivery
The rate of neonatal malformations and developmental disorders | 1-2 days after delivery
birth weight | At delivery
Head circumference | 1-2 days after delivery
Maternal adverse effects | During the length of pregnancy (up to 9 months)
Duration of time until pharmacotherapy for glycemic control is indicated | During the length of pregnancy (up to 9 months)

CONTACTS AND LOCATIONS:
Locations (4):
- Israel (4):
  - Assuta-Ashdod medical center, Ashdod
  - Rambam medical center, Haifa
  - Wolfson medical center, Holon
  - Poriya Medical center, Tiberias

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nachum Z, Perlitz Y, Shavit LY, Magril G, Vitner D, Zipori Y, Weiner E, Alon AS, Ganor-Paz Y, Nezer M, Harel N, Soltsman S, Yefet E. The effect of oral probiotics on glycemic control of women with gestational diabetes mellitus-a multicenter, randomized, double-blind, placebo-controlled trial. Am J Obstet Gynecol MFM. 2024 Jan;6(1):101224. doi: 10.1016/j.ajogmf.2023.101224. Epub 2023 Nov 12. PMID 37956906
- [Derived] Okesene-Gafa KA, Moore AE, Jordan V, McCowan L, Crowther CA. Probiotic treatment for women with gestational diabetes to improve maternal and infant health and well-being. Cochrane Database Syst Rev. 2020 Jun 24;6(6):CD012970. doi: 10.1002/14651858.CD012970.pub2. PMID 32575163